CLINICAL TRIAL: NCT00004207
Title: A Phase I Study to Determine the Maximum Tolerated Dose of Daunoxome as Therapy for the Treatment of Metastatic Breast Cancer
Brief Title: Liposomal Daunorubicin in Treating Patients With Metastatic Breast Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Leicester (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067453; LRI-103-UK-V1.1; EU-99033
Record Dates: First submitted 2000-01-21; First posted 2004-08-09 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2000-07

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Daunorubicin

INTERVENTIONS:
Drug: liposomal daunorubicin citrate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of liposomal daunorubicin in treating patients who have metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of daunorubicin liposomal in patients with metastatic breast cancer. II. Assess the antineoplastic activity and safety profile of this regimen in these patients.

OUTLINE: This is a dose escalation study. Patients receive daunorubicin liposomal IV over a minimum of 2 hours on day 1. Treatment repeats every 3 weeks for a maximum of 8 courses in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of daunorubicin liposomal until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 2 of 6 patients experience dose limiting toxicity. Patients with stable or responding disease are followed at 1 and 3 months, then every 3 months for 1 year.

PROJECTED ACCRUAL: Approximately 15-20 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically proven metastatic breast cancer Measurable disease No bone metastases only No CNS involvement or leptomeningeal disease Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: 18 and over Menopausal status: Not specified Performance status: ECOG 0-2 Life expectancy: At least 3 months Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 9 g/dL Hepatic: Bilirubin less than 1.5 times upper limit of normal (ULN) AST or ALT less than 2 times ULN (less than 5 times ULN if liver metastases present) Renal: Creatinine normal Cardiovascular: Left ventricular ejection fraction at least 50% or normal by echocardiogram or MUGA scan No active ischemic heart disease No uncontrolled hypertension No poorly controlled atrial arrhythmias, symptomatic angina pectoris, or myocardial infarction within the past 6 months No symptomatic congestive heart failure, percutaneous transluminal coronary angioplasty, or coronary artery bypass graft surgery within the past 12 months Other: No other primary cancer within the past 5 years except curatively treated nonmelanomatous skin cancer or carcinoma in situ of the cervix Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No condition that would preclude informed consent or compliance

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 3 weeks since prior immunotherapy No prior bone marrow transplantation Chemotherapy: Prior nonanthracycline based chemotherapy for breast cancer allowed No prior anthracycline based chemotherapy for metastatic disease Prior anthracycline based adjuvant chemotherapy allowed if: At least 6 months have elapsed from completion of adjuvant therapy until the detection of metastatic disease Cumulative dose no greater than 300 mg/m2 Endocrine therapy: At least 3 weeks since prior hormonal therapy No concurrent hormonal or corticosteroid therapy for breast cancer Radiotherapy: At least 2 weeks since prior radiotherapy and recovered No concurrent radiotherapy Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1997-12

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth O'Byrne, MD, Study Chair — University Hospitals, Leicester
Locations (1):
- Leicester Royal Infirmary NHS Trust, Leicester, England, United Kingdom